CLINICAL TRIAL: NCT07088107
Title: Development and Validation of an Adaptive Neurofeedback Interface Using Transcranial Magnetic Stimulation to Modulate Cortical Excitability
Brief Title: A Neurofeedback Interface in Poststroke Neuromodulation Using TMS-fNIRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HSEARS20240902001
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Neurofeedback; Brain Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- functional near-infrared spectroscopy (fNIRS)-triggered TMS (Experimental): The TMS will be triggered based on individualized fNIRS signals from the participants. Specifically, the TMS will be triggered during ascending phase of fNIRS hemodynamic response during motor imagination.
  Interventions: Device: fNIRS-triggered TMS
- Sham functional near-infrared spectroscopy (fNIRS)-triggered TMS (Sham Comparator): The TMS will be triggered by fNIRS obtained by another participant.
  Interventions: Device: fNIRS-triggered TMS

INTERVENTIONS:
Device: fNIRS-triggered TMS — The firing of TMS will be triggered according to fNIRS signal intensity.

SUMMARY:
Stroke is a type of cerebrovascular disease, and the primary characteristic of post-stroke brains is pathological changes in cerebral hemodynamics. Therefore, hemodynamic signals may provide straightforward information for guiding post-stroke neuromodulation therapy. Transcranial magnetic stimulation (TMS), a non-invasive neurostimulation modality, has been extensively used in post-stroke rehabilitation. However, current TMS-based neuromodulation therapy demonstrates a large treatment response variability due to its open-loop nature. To address this challenge, the research team will develop a novel form of closed-loop neurofeedback interfaces which controls the timing of TMS pulses precisely based on neural biomarkers from functional near-infrared spectroscopy (fNIRS) and test the accuracy of the adaptive neurofeedback system in healthy adults. After establishing the TMS-based neurofeedback interface, a proof-of-concept study enrolling postacute stroke patients will be performed to evaluate the efficacy of the TMS neurofeedback interface in enhancing motor control of the hemiplegic upper extremity and cortical excitability of the ipsilesional motor cortex. These findings will verify whether the proposed fNIRS-controlled TMS neurofeedback interface can be clinically feasible as a form of post-stroke neuromodulation therapy. Additionally, the results will significantly contribute to the scientific understanding of how neuromodulation improves hemodynamic signals in a closed-loop manner, thereby enhancing functional recovery in poststroke survivors.

DETAILED DESCRIPTION:
Stroke is a type of cerebrovascular disease, and the primary characteristic of post-stroke brains is pathological changes in cerebral hemodynamics. Therefore, hemodynamic signals may provide straightforward information for guiding post-stroke neuromodulation therapy. Transcranial magnetic stimulation (TMS), a non-invasive neurostimulation modality, has been extensively used in post-stroke rehabilitation. However, current TMS-based neuromodulation therapy demonstrates a large treatment response variability due to its open-loop nature. To address this challenge, the research team will develop a novel form of closed-loop neurofeedback interfaces which controls the timing of TMS pulses precisely based on neural biomarkers from functional near-infrared spectroscopy (fNIRS) and test the accuracy of the adaptive neurofeedback system in healthy adults. After establishing the TMS-based neurofeedback interface, a proof-of-concept study enrolling postacute stroke patients will be performed to evaluate the efficacy of the TMS neurofeedback interface in enhancing motor control of the hemiplegic upper extremity and cortical excitability of the ipsilesional motor cortex. These findings will verify whether the proposed fNIRS-controlled TMS neurofeedback interface can be clinically feasible as a form of post-stroke neuromodulation therapy. Additionally, the results will significantly contribute to the scientific understanding of how neuromodulation improves hemodynamic signals in a closed-loop manner, thereby enhancing functional recovery in poststroke survivors.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet the following criteria will be included:

1. Diagnosed with ischemic subcortical stroke, with stroke onset≥6 months.
2. Age between 18 and 80 years.
3. Residual upper limb functions between levels 2-7 in the FTHUE.
4. Capable of providing informed written consent.
5. Capable of reading and communicating with Chinese.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded:

1. any contraindications to TMS (screened by the safety checklist by Rossi).
2. Diagnosed with any concomitant neurological disease other than stroke.
3. signs of cognitive impairment, with a Montreal cognitive assessment score<21/22 out of 30.
4. Severe spasticity in the hemiparetic upper limb muscles, with a Modified Ashworth score > 2.
5. any moderate-to-severe chronic illness, such as uncontrolled hypertension, heart disease or renal failure.

Healthy participants should be aged between 18 and 80, with no known history of neurological diseases. They should not have any moderate-to-severe chronic illness, such as uncontrolled hypertension, heart disease or renal failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potential | Baseline
  Motor Evoked Potentials (MEPs) are electrical signals generated by stimulating the motor cortex and recorded from the peripheral muscle (e.g., a hand muscle). This is a measure of corticospinal excitability.
Motor Evoked Potentials (MEPs) | After 1 hour
  Motor Evoked Potentials (MEPs) are electrical signals generated by stimulating the motor cortex and recorded from the peripheral muscle (e.g., a hand muscle). This is a measure of corticospinal excitability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided